CLINICAL TRIAL: NCT03311828
Title: A Pilot/Feasibility Trial of 64Cu-DOTA-Daratumumab Positron Emission Tomography in Patients With Newly Diagnosed or Relapsed Multiple Myeloma
Brief Title: Copper 64Cu-DOTA-Daratumumab Positron Emission Tomography in Diagnosing Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17141; NCI-2017-01873 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Plasma Cell Myeloma; Plasma Cell Myeloma; Secondary Amyloidosis
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Copper 64Cu-DOTA-daratumumab, PET) (Experimental): Patients receive daratumumab IV over 10-45 minutes, and within 6 hours, patients receive copper 64Cu-DOTA-daratumumab IV on day 0. Patients undergo PET on days 1 and 2.
  Interventions: Biological: Daratumumab; Drug: Imaging Agent; Procedure: Positron Emission Tomography; Other: Pharmacological Study

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: 945721-28-8; Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Imaging Agent — Given Copper 64Cu-DOTA-daratumumab IV
  Other Names: Image Enhancement Agent
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging; PET; PET Scan; positron emission tomography scan; proton magnetic resonance spectroscopic imaging
Other: Pharmacological Study — Correlative studies

SUMMARY:
This pilot phase I clinical trial studies how well copper 64Cu-DOTA-daratumumab positron emission tomography works in diagnosing patients with multiple myeloma that has come back. Diagnostic procedures, such as copper 64Cu-DOTA-daratumumab positron emission tomography, may help evaluate the extent of multiple myeloma in patients prior to the initiation of treatment and ultimately monitor disease status/response during and post treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety and tolerability of unlabeled daratumumab followed by 64Cu-DOTA-daratumumab positron emission tomography, at each dose level, by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. Generate initial estimates of the biodistribution of the 64Cu-DOTA-daratumumab and the preferred dose of cold antibody.

II. Determine the dose of pre-administered unlabeled daratumumab that optimizes image quality of 64Cu-anti-CD38 (daratumumab)-NHS-DOTA.

III. Evaluate the sensitivity of 64Cu-anti-CD38 (daratumumab)-NHS-DOTA in detecting lesions compared to 18F fludeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) scanning.

OUTLINE:

Patients receive daratumumab intravenously (IV) over 10-45 minutes, and within 6 hours, patients receive copper 64Cu-DOTA-daratumumab IV on day 0. Patients undergo PET on days 1 and 2.

After completion of study, patients are followed up for 7 days and then at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Histologically confirmed multiple myeloma (newly diagnosed or relapsed)(Note: multiple myeloma patients with secondary amyloidosis are eligible)
* Ability to undergo standard PET imaging; an 18 F FDG PET/CT scan will take place within 3 months of enrollment
* Karnofsky performance status > 70%
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 50/mm^3; platelet transfusions to help patients meet eligibility criteria are not allowed within 7 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30 mL/min
* Woman of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods; condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization; true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (6 months after the last dose of 64 Cu-anti-CD38 [daratumumab]-NHS-DOTA for women)

  * A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 6 months after receiving the last dose of study drug

Exclusion Criteria:

* Daratumumab or other anti CD38 antibody treatment within 3 months prior to study enrollment
* Female patients who are lactating or have a positive pregnancy test during the screening period
* Major surgery within 14 days prior to start of study treatment
* Infection requiring systemic antibiotic therapy within 14 days prior to start of study treatment
* Subject is receiving concurrent chemotherapy or biologic or hormonal therapy for cancer treatment; subject is receiving bone marrow stimulatory factors (e.g., granulocyte-macrophage colony-stimulating factor [GM-CSF]); Note: Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes) is acceptable
* Vaccination with live attenuated vaccines within 4 weeks of study agent administration
* Subject is currently using or has used immunosuppressive medication within 14 days prior to the study agent administration; the following are exceptions:

  * Intranasal, topical, inhaled, or local steroid injections (e.g., intra-articular injection)
  * Chronic systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., infusion-related reactions, CT scan premedication)
* Subject has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloidosis
* Subject has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% predicted normal; Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 < 50%
* Subject has known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or investigator's brochure)
* Subject has history of primary immunodeficiency
* Subject is positive for human immunodeficiency virus (HIV-1), chronic or active hepatitis B, or active hepatitis A or C
* Subject has any one of the following:

  * Clinically significant abnormal electrocardiography (ECG) finding at screening
  * Congestive heart failure (New York Heart Association class III or IV)
  * Myocardial infarction within 12 months prior to starting study treatment
  * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
* Subject has presence of other active malignancy (see exceptions below) (However, research participants with history of prior malignancy treated with curative intent and in complete remission are eligible). The following malignancies are exceptions to the active malignancy statement:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM clinical staging system) or prostate cancer that is curative
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event | Up to 7 days
  Will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03. Observed toxicities will be summarized, for all dose levels, in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study agent(s) and reversibility or outcome.

SECONDARY OUTCOMES:
Detection of lesions in the body | Up to 7 days
  Will be determined by copper 64Cu-DOTA-daratumumab positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Krishnan A, Adhikarla V, Poku EK, Palmer J, Chaudhry A, Biglang-Awa VE, Bowles N, Nathwani N, Rosenzweig M, Sahebi F, Karanes C, Simpson J, Sanchez JF, Yamauchi D, Parayno M, Chowdhury A, Caserta E, Marcucci G, Rockne R, Wu AM, Wong J, Forman SJ, Colcher D, Yazaki P, Shively J, Pichiorri F. Identifying CD38+ cells in patients with multiple myeloma: first-in-human imaging using copper-64-labeled daratumumab. Blood Adv. 2020 Oct 27;4(20):5194-5202. doi: 10.1182/bloodadvances.2020002603. PMID 33095874